CLINICAL TRIAL: NCT02878902
Title: Impact of the Implementation of a Chronic Kidney Disease (CKD) Coordination Function on Dialysis Initiation Frequency in Emergency
Brief Title: Impact of the Implementation of CKD Coordination Function on Dialysis Initiation Frequency in Emergency
Acronym: ICoDU
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 15-199
Record Dates: First submitted 2016-07-29; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Kidney Disease
Keywords: emergency; coordination; dialysis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Before implementation: Patients registered in monitoring French registry of renal patients "Réseau Epidémiologie et Information en Néphrologie" (REIN) from January 1, 2012 to December 31, 2013
- Post implementation: Patients registered in monitoring French registry of renal patients "Réseau Epidémiologie et Information en Néphrologie" (REIN) from January 1, 2014 to December 31, 2015
  Interventions: Other: Post implementation

INTERVENTIONS:
Other: Post implementation — Patient group whose care course was organized by the nurse coordinator of chronic renal failure
  Groups: Post implementation

SUMMARY:
Kidney failure is a major public health problem. REIN registry shows that 33% of patients treated in renal replacement therapy for ESRD start dialysis in emergency. Unscheduled care is associated with an increased risk of morbidity and mortality, with less access to off dialysis center and kidney transplant. In addition, the emergency management has an impact on the organization of health structures. The High Authority of Health in 2012 issued a "care pathway Guide" aimed "to report in this process of the multidisciplinary nature of the management and coordination of principles and procedures for the Chronic Renal failure and cooperation between professionals involved. " A function of coordinator of the Chronic Renal Disease was set up in service since May 2013. Investigators propose to carry out a study to value its impact on the start of the dialysis in emergency and hypothesize that this feature innovative in France improves the patient pathway and thus reduce support emergency frequency of ESRD.

The objective of this study is to show the improvement of the quality of care for terminally chronic renal failure patients.

This is to evaluate an experiment aimed to facilitate a complex care path. If this experiment is successful, it could form part of "advanced practice".

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with terminal chronic renal failure enrolled in the course of care

Exclusion Criteria:

* Patients under 18 years
* Patient Off Course
* Patient beginning dialysis with a method of transition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with chronic kidney disease in our center
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of emergency dialysis patients beginner | Change of this percentage from baseline at 2 years
  The outcome is mesured at baseline (implementation of the nurse coordinator of chronic renal failure
  the nurse coordinator of chronic renal failure
  Baseline = implementation of this function of coordination of patients with chronic renal failure

IPD SHARING:
Plan to Share IPD: No